CLINICAL TRIAL: NCT03645395
Title: A Phase 2a Open-label Study to Investigate Safety and Tolerability (Including the Maximum Tolerated Dose), Efficacy, Pharmacokinetics, Pharmacodynamics and Immunogenicity of MT-3724 in Combination With Lenalidomide in Subjects With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Multiple Dose Regimens of MT-3724 With Lenalidomide for the Treatment of Participants With Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma (MT-3724_NHL_003)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Molecular Templates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MT-3724_NHL_003
Record Dates: First submitted 2018-07-19; First posted 2018-08-24 (Actual); Results first posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Non-hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MT-3724 10 mcg/kg-LEN (Experimental): MT-3724 10 mcg/kg/dose IV for 6 doses over 12 days (M-W-F X 2 weeks on Days 1, 3, 5, 8, 10, and 12) of each 28 day cycle in combination with LEN. If the treatment with MT-3724 is continued beyond Cycle 2, then MT-3724 will be administered weekly (Days 1, 3, 5, 8, 10, and 12) of each 28-day cycle
  Interventions: Drug: MT-3724
- MT-3724 25 mcg/kg-LEN 3x a week (Experimental): MT-3724 25 mcg/kg/dose IV for 6 doses over 12 days (M-W-F X 2 weeks on Days 1, 3, 5, 8, 10, and 12) of each 28 day cycle in combination with LEN. If the treatment with MT-3724 is continued beyond Cycle 2, then MT-3724 will be administered weekly Days 1, 3, 5, 8, 10, and 12) of each 28-day cycle
  Interventions: Drug: MT-3724
- MT-3724 20 mcg/kg-LEN 3x a week (Experimental): MT-3724 20 mcg/kg/dose IV for 6 doses over 12 days (M-W-F X 2 weeks on Days 1, 3, 5, 8, 10, and 12) of each 28 day cycle in combination with LEN. If the treatment with MT-3724 is continued beyond Cycle 2 , then MT-3724 will be administered weekly (Days 1, 3, 5, 8, 10, and 12) of each 28-day cycle
  Interventions: Drug: MT-3724
- MT-3724 25 mcg/kg-LEN 2x a week (Experimental): MT-3724 25 mcg/kg dose IV for 4 doses (days 1, 5, 8 and 12 during cycles 1 and 2) of each 28 day cycle in combination with LEN and weekly during cycles 3 and beyond (days 1, 8, 15 and 22).
  Interventions: Drug: MT-3724
- MT-3724 50 mcg/kg-LEN (Experimental): MT-3724 50 mcg/kg dose IV for 4 doses (days 1, 5, 8 and 12 during cycles 1 and 2) of each 28 day cycle in combination with LEN and weekly during cycles 3 and beyond (days 1, 8, 15 and 22).
  Interventions: Drug: MT-3724

INTERVENTIONS:
Drug: MT-3724 — Experimental treatment with MT-3724 in combination with LEN therapy.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of MT-3724 in combination with Lenalidomide in participants with relapsed or refractory B-Cell NHL.

DETAILED DESCRIPTION:
This is a multi-center, open-label two-part study evaluating the safety and tolerability of MT-3724 in combination with Lenalidomide in relapsed or refractory CD20 positive B-cell Lymphoma participants.

Part 1: (MT-3724 Dose Escalation) Define the maximum tolerated dose (MTD) of MT-3724 in combination with standard treatment of Lenalidomide

Part 2: (MTD Expansion Cohort) Confirm the safety and tolerability of the MTD of MT-3724 from Part 1 in the MTD Expansion Cohort, where MT-3724 will be given at the MTD in combination with Lenalidomide. In addition, the Pharmacokinetics (PK), Pharmacodynamics (PD), immunogenicity and tumor response at the MTD of MT-3724 in combination with Lenalidomide will be more thoroughly evaluated in Part 2.

It is anticipated that up to 64 participants will be enrolled. Treatment will continue until disease progression, withdrawal of consent or any other reason.

ELIGIBILITY:
Inclusion Criteria:

- Participants must meet ALL the following criteria to be eligible for the study.

1. Be adequately informed about the study and fully consent to participation as demonstrated by signing the written ICF before any screening procedure.
2. Be aged ≥18 years years on the date of signing the informed consent form.
3. Have relapsed or refractory CD20 positive B-cell NHL that, in the investigator's opinion, could benefit from MT-3724+LEN therapy. Participants must have proof of CD20 positive NHL either by:

   1. Historical biopsies (obtained with diagnosis of relapsed or refractory disease), or
   2. Fresh biopsies.

      * Bone marrow biopsy
      * Excisional lymph node biopsy
   3. Core biopsy of any involved organ; all are acceptable methods; FNA not acceptable
4. All subtypes of B-cell NHL may be considered for Part 1 (MT-3724 dose escalation). Only histologically documented DLBCL (including mixed histology) may be considered for Part 2 (MTD expansion cohort).
5. Have received all available approved therapies for NHL, one of which should be anti-CD20 based therapy.

   1. Participants whose prior therapy includes chimeric antigen receptor t-cell (CAR-T) cell therapy are eligible.
   2. Participants who underwent stem cell transplant (SCT) >100 days for autologous SCT or >180 days for allogeneic SCT before study drug administration and exhibited a full hematological recovery (consistent with the existing inclusion criteria requirements and without PRBC or platelet transfusions within 2 weeks of C1D1) prior to relapse are eligible.
6. Have bi-dimensionally measurable disease by Lugano Classification for NHL:

   1. >1.5 cm LDi for lymph nodes
   2. >1.0 cm LDi for extra nodal disease.
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2
8. Have adequate bone marrow function, as determined by all the following:

   1. Absolute neutrophil count (ANC) ≥1,000/mm³
   2. Platelet count ≥50,000 mm³
   3. Hemoglobin ≥8g/dL
9. Have adequate kidney function, creatinine clearance (CLcr) to be ≥50mL/min either measured or assessed by using the Cockcroft-Gault formula.

   a. At the investigator's discretion, the eGFR result ≤50 mL/min may be verified by measurement of CLcr based on the 24-hour urine collection. Participants with CLcr ≥50 mL/min will be eligible irrespective of the eGFR result.
10. Have adequate hepatic function, as determined by:

    1. Total bilirubin ≤1.5 x upper limit normal (ULN), or direct bilirubin ≤1.5 x ULN for participants with elevated total bilirubin secondary to Gilbert's Syndrome) and
    2. Aspartate aminotransferase (AST) ≤3 x ULN (or ≤5 x ULN if liver involvement) and
    3. Alanine aminotransferase (ALT) ≤3 x ULN (or ≤5 x ULN if liver involvement)
11. Have adequate coagulation, as determined by:

    1. International Normalized Ration (INR) or Prothrombin Time (PT) ≤1.5 x ULN (unless on therapeutic anticoagulants)
    2. Activated partial thromboplastin time (aPTT) ≤1.5 x ULN (unless on therapeutic anticoagulants)
12. Albumin ≥ 3.0 g/dL
13. Women of reproductive potential must have a negative pregnancy test on 2 occasions during the screening period (within 10-14 days and within 24 hours before the start of treatment). Women not of reproductive potential are female participants who are postmenopausal(>1 year since last menstrual cycle) or permanently sterilized (e.g., hysterectomy, bilateral salpingectomy).
14. Males must agree to always use a latex or synthetic condom during any sexual contact with females of reproductive potential while taking LEN and for up to 4 weeks after discontinuing LEN, even if they have undergone a successful vasectomy. Male participants taking LEN must not donate sperm.
15. Participants of reproductive potential and their partners must agree to either to abstain continuously from heterosexual intercourse or to use 2 methods of reliable birth control simultaneously to begin 4 weeks prior to initiating treatment with LEN until 28 days after the last dose of MT-3724 or LEN. The investigator or a designated associate should advise the participants how to achieve adequate contraception. The following birth control methods may be considered: one highly effective form of contraception - tubal ligation, intrauterine device (IUD), hormonal (birth control pills, injections, hormonal patches, vaginal rings, or implants), or partner's vasectomy, and one additional effective contraceptive method - male latex or synthetic condom, diaphragm, or cervical cap.
16. Participants must have a life expectancy of >3 months from the start of treatment.

Exclusion Criteria:

* Participants who meet any of the following criteria must be excluded from the study.

Medical and surgical history

1. History or current evidence of neoplastic disease that is histologically distinct from NHL, except cervical carcinoma in situ, superficial noninvasive bladder tumors, curatively treated Stage I-II non-melanoma skin cancer. Participants with prior, curatively treated cancer >2 years ago before the start of treatment can be enrolled.
2. Current evidence of new or growing brain or spinal metastases during screening. Participants with known brain or spinal metastases may be eligible if they:

   1. Had radiotherapy or another appropriate therapy for the brain or spinal metastases; concurrent prophylactic treatment is allowed.
   2. Neurological symptoms must be stable and no worse than grade 2
   3. Have evidence of stable brain or spinal disease on computer topography (CT) or magnetic resonance imaging (MRI) scan obtained within 4 weeks of signing the ICF and compared with prior imaging results.
   4. Do not require chronic steroid therapy, or if applicable, have been stable on steroid dose of no more than prednisone 20mg/day or equivalent by C1D1.
3. Current evidence of Graft versus Host Disease.
4. Current evidence of Common Terminology Criteria for Adverse Events (CTCAE) Grade >1 toxicity (before the start of treatment, except for hair loss, and those Grade 2 toxicities listed as permitted in other eligibility criteria).
5. Current evidence of incomplete recovery from surgery or radiotherapy before the start of treatment, or planned surgery or radiotherapy at any time during the study until the EoT Visit, except minor elective interventions deemed acceptable by the investigator.
6. Current evidence of significant (CTCAE Grade ≥2) infection or wound within 4 weeks before the start of treatment.

   a. Participants with Grade 2 infection that has stabilized or improved with oral anti-infectives before the start of treatment may be eligible at the sponsor's discretion
7. Current evidence of significant cardiovascular disease including, but not limited to the following conditions:

   1. Unstable angina (symptoms of angina at rest) or new-onset angina within ≤3 months before the start of treatment.
   2. Arterial thrombosis or pulmonary embolism within ≤3 months before the start of treatment.
   3. Myocardial infarction or stroke within ≤3 months before the start of treatment.
   4. Pericarditis (any CTCAE grade), pericardial effusion (CTCAE Grade ≥2), non malignant pleural effusion (CTCAE Grade ≥2) or malignant pleural effusion (CTCAE Grade ≥3).
   5. Congestive heart failure New York Heart Association (NYHA) Class III or IV at screening or left ventricular ejection fraction (LVEF) <45%, assessed by Echo or multiple-gated acquisition (MUGA) scan within 1 month before starting study treatment. (inclusion of participants with LVEF between 40%-45% should be discussed and approved by the sponsor). Echo or MUGA scan performed within 6 months before screening and at least 28 days after the last cancer therapy is acceptable provided the participant has not received any potential cardiotoxic agents since then.
   6. Cardiac arrhythmia requiring anti-arrhythmic therapy at Screening. Participants receiving digoxin, calcium channel blockers, or beta-adrenergic blockers are eligible at the investigator's discretion after consultation with medical monitor if the dose has been stable for ≥2 weeks before the start of treatment with MT-3724. Participants with sinus arrhythmia and infrequent premature ventricular contractions are eligible at the investigator's discretion.
8. QT interval corrected according to Fridericia's formula (QTcF) >480 ms, determined as the average from three QTcF values on the triplicate electrocardiogram (ECG) obtained at Screening.
9. Current evidence of uncontrolled HIV, HBV or HCV at screening. Serology testing is not required if seronegativity is documented in the medical history and if there are no clinical signs suggestive of HIV or hepatitis infections, or suspected exposure. The following exceptions apply for participants with positive viral serology:

   1. Participants with HIV and an undetectable viral load and CD4+ T-cells counts ≥350 cells/microliter may be enrolled, but must be taking appropriate opportunistic infection prophylaxis, if clinically relevant.
   2. Participants with positive HBV serology are eligible if they have an undetectable viral load and the participant will receive antiviral prophylaxis for potential HBV reactivation-per institutional guidelines.
   3. Participants with positive HCV serology are eligible if quantitative PCR for plasma HCV RNA is below the lower limit of detection. Concurrent antiviral HCV treatment per institutional guidelines is allowed.
10. Women who are pregnant or breastfeeding.
11. History or current evidence of hypersensitivity to any of the study drugs, or of current hypersensitivity requiring systemic steroids at doses >20 mg/day prednisone equivalent.
12. History or current evidence of any other medical or psychiatric condition or addictive disorder, or laboratory abnormality that, in the opinion of the investigator, may increase the risks associated with study participation, or require treatments that may interfere with the conduct of the study or the interpretation of study results.

    Prior treatments
13. Prior treatment with MT-3724.
14. Received anti-CD20 monoclonal antibody (Mab) therapy within the following periods before the start of treatment

    1. Rituximab (Rituxan® RTX): 84 days; if a participant had received RTX within 37 Weeks before the start of treatment, then a serum RTX level must be negative (<500 ng/mL) at screening.
    2. Obinutuzumab (Gazyva®): 184 days
    3. Ofatumumab (Arzerra®): 88 days
15. Received therapy for NHL (except the anti-CD20 Mab therapies listed above and radioimmunoconjugates) within 4 weeks before the start of treatment.
16. Any investigational drug treatment from 4 weeks or 5 half-lives of the agent before the start of treatment, whichever is longer, until the EoT Visit.
17. Received radiotherapy to tumor lesions that would be chosen as target lesions (measurable disease) within 4 weeks before the start of treatment, unless the lesion exhibited objective progression between the radiotherapy and the screening according to the Lugano Classification for NHL.

    a. Palliative radiotherapy to non-target lesions may be permitted at the investigator's discretion after consultation with the medical monitor.
18. Received any live vaccines within 4 weeks before of the start of treatment, unless the investigator believes the benefits outweigh the risks, after approval with the sponsor.
19. Require use of systemic immune modulators during study treatment. a. Systemic immune modulators include but are not limited to systemic corticosteroids at doses >20 mg/day or prednisone equivalent, cyclosporine and tacrolimus.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Innovative Clinical Research Institute, Whittier, California
  - Boca Raton Clinical Research, Plantation, Florida
  - Rush University, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This two-part [Part 1: Dose Escalation and Part 2: maximum tolerated dose (MTD) Expansion Cohort] study evaluated the safety and tolerability of MT-3724 in combination with Lenalidomide (LEN) in participants with relapsed or refractory CD20 positive B-cell Lymphoma.
Pre-assignment Details: Total 9 participants were enrolled in the study. Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Groups:
- Part 1: MT-3724 10 mcg/Kg-LEN: Participants were administered MT-3724 10 micrograms per kilograms/dose intravenously (mcg/kg/dose IV) on Days 1,3,5,8, 10 and 12 on Cycle 1 and 2 and Cycle 3 onwards Days 1,8,15 and 22. Participants self-administered 20 mg LEN on the first 21 consecutive days (D1-D21) of each 28-day cycle.
- Part 1: MT-3724 25 mcg/Kg-LEN: Participants were administered MT-3724 25 mcg/kg/dose IV on Days 1,3,5,8, 10 and 12 on Cycle 1 and 2 and Cycle 3 onwards Days 1,8,15 and 22. Participants self-administered 20 mg LEN on the first 21 consecutive days (D1-D21) of each 28-day cycle.
- Part 1: MT-3724 20 mcg/Kg-LEN: Participants were administered MT-3724 20 mcg/kg/dose IV on Days 1,3,5,8, 10 and 12 on Cycle 1 and 2 and Cycle 3 onwards Days 1,8,15 and 22. Participants self-administered 20 mg LEN on the first 21 consecutive days (D1-D21) of each 28-day cycle.
- Part 2: MT-3724 50mcg/Kg-LEN: Participants were to be administered MT-3724 50 mcg/kg/dose IV on Days 1,3,5,8, 10 and 12 on Cycle 1 and 2 and Cycle 3 onwards Days 1,8,15 and 22. Participants were to self-administer 20 mg LEN on the first 21 consecutive days (D1-D21) of each 28-day cycle.
Period: Part 1 (Up to 6 Months)
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Started | 3 | 3 | 3 | 0
Completed | 1 | 0 | 0 | 0
Not Completed | 2 | 3 | 3 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Sponsor's decision to close the trial | 1 | 2 | 2 | 0
Period: Part 2 (Up to 6 Months)
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Groups:
- Part 1: MT-3724 10 mcg/Kg-LEN: Participants were administered MT-3724 10 mcg/kg/dose IV on Days 1,3,5,8, 10 and 12 on Cycle 1 and 2 and Cycle 3 onwards Days 1,8,15 and 22. Participants self-administered 20 mg LEN on the first 21 consecutive days (D1-D21) of each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN | Total
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (8.33) | 61.3 (8.33) | 71.0 (12.77) |  | 64.9 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 |  | 6
  Male | 0 | 2 | 1 |  | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 1 | 1 |  | 3
  White | 2 | 2 | 1 |  | 5
  Other | 0 | 0 | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1 and 2: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious AEs (SAEs) and Dose-limiting Toxicity
Description: An adverse event is any untoward medical occurrence or clinical investigation in a participant administered a pharmaceutical product(s) and which does not necessarily have to have a causal relationship with this experimental treatment(s). SAE is any untoward medical occurrence, at any dose; is fatal or life-threatening, is life-threatening, results in permanently disabling; results in unplanned in-patient hospitalization or prolongation of existing hospitalization; results in a congenital abnormality or birth defect; important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when based upon appropriate medical judgment, they may jeopardize the participant or may require medical or surgical intervention. A DLT is any TEAE that occurred after the start of infusion in cycle 1 of Part 1 and the TEAE is at least possibly related to the study drug, as determined by the sponsor after consultation with the investigator(s).
Time Frame: Up to 1 year
Population: Safety Population included participants who received at least one dose of any study drug (either MT-3724, or lenalidomide). Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Measure: Number; unit: participants
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 3 | 3 | 3 | 0
participants
  TEAEs | 3 | 3 | 3 |
  SAEs | 1 | 1 | 1 |
  DLT | 0 | 2 | 0 |

2. Primary Outcome: Part 1 and 2: Number of Participants With Abnormal Laboratory Parameters
Description: Laboratory parameters included hematology, blood chemistry, and urinalysis. Any abnormal laboratory test results which were considered clinically significant by the investigator were recorded on the case report form. Number of participants with any clinically significant abnormalities in laboratory parameters have been presented.
Time Frame: Up to 1 year
Population: Safety Population. Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Measure: Number; unit: Participants
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 3 | 3 | 3 | 0
Participants | 3 | 3 | 3 |

3. Primary Outcome: Part 1 and 2: Number of Participants With Clinically Significant Physical Findings
Description: This analysis was planned but data was not captured in the database. Abnormal changes were captured as adverse events if they were clinically significant.
Time Frame: Up to 1 year
Population: Safety population. Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Part 1 and 2: Plasma Concentrations of MT-3724
Description: Blood samples were collected for Pharmacokinetic (PK) analysis of MT-3724. Data could not be calculated due to small sample size and inconsistent sampling as a result of early termination.
Time Frame: Days 1,3 and 12 of treatment cycle (Each cycle is of 28 days); Up to 1 year
Population: PK population included all participants who received at least one dose of MT-3724 and have at least one post-baseline PK assessment. Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 3 | 3 | 3 | 0
Micrograms per milliliter | NA (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) | NA (NA) — Mean and Standard Deviation could not be calculated due to high proportion of non-quantifiable values (>30 percent [%] of values were imputed) |

5. Secondary Outcome: Part 1 and 2: Change From Baseline in B-cell Count
Description: Blood samples were collected for analysis of B-cell count. Data could not be calculated due to small sample size and inconsistent sampling as a result of early termination.
Time Frame: Up to 1 year
Population: Pharmacodynamic (PD) Population included all participants who received at least one dose of MT-3724 and have at least one post-baseline PD assessment. Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 3 | 3 | 3 | 0
Giga cells per liter | NA (NA) — Mean and Standard Deviation could not be calculated as 100% of the data was below the limit of quantification at all time points. | NA (NA) — Mean and Standard Deviation could not be calculated as 100% of the data was below the limit of quantification at all time points. | NA (NA) — Mean and Standard Deviation could not be calculated as 100% of the data was below the limit of quantification at all time points. |

6. Secondary Outcome: Part 1 and 2: Number of Participants With Anti-drug Antibody Titer When Treated With MT-3724
Description: Blood samples were collected for analysis of ADA titer. Data was not collected due to early termination of the trial.
Time Frame: Up to 1 year
Population: Immunogenicity Population included all participants who received at least one dose of MT-3724 and have at least one post-baseline immunogenicity assessment. Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Part 1 and 2: Number of Participants With Neutralizing Antibody (NAb) Titers When Treated With MT-3724
Description: Blood samples were planed to be collected for analysis of neutralizing antibody (NAb) titers. Data was not collected due to early termination of the trial.
Time Frame: Up to 1 year
Population: as for outcome 6
Groups:
- Part 2: MT-3724 50mcg/Kg-LEN: Participants were to be administered MT-3724 50 mcg/kg/dose IV on Days 1,3,5,8, 10 and 12 on Cycle 1 and 2 and Cycle 3 onwards Days 1,8,15 and 22. Participants to self-administer 20 mg LEN on the first 21 consecutive days (D1-D21) of each 28-day cycle.
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Part 1 and 2: Number of Participants With Objective Response Rate (ORR)
Description: ORR was defined as CR or Partial Response (PR). CR: a score 1 (no uptake above background), 2 (uptake <=mediastinum), or 3 (<mediastinum but <=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites with no new lesions and no evidence of FDG-avid disease in bone marrow. PR: a score 4 (uptake moderately greater than [>] liver) or 5 (uptake markedly >liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size on PET 5-PS for lymph nodes and extralymphatic sites with no new lesions and reduced residual uptake in bone marrow compared with baseline. Higher score indicates worse outcomes.
Time Frame: Up to 1 year
Population: Safety population. Part 2 was not initiated due to Sponsor's decision to terminate the trial. The rows presenting data for PR and CR are mutually exclusive.
Measure: Number; unit: participants
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 3 | 3 | 3 | 0
participants
  PR | 2 | 0 | 1 |
  CR | 1 | 2 | 1 |

9. Secondary Outcome: Part 1 and 2: Duration of Response (DOR)
Description: DOR is defined as the time from the first documented complete or partial response to the actual date of disease progression or death before progression. Data was not collected due to early termination of the trial.
Time Frame: Up to 1 year
Population: Safety population. Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Part 1 and 2: Progression Free Survival (PFS)
Description: PFS is defined as the time from first dose date until the first occurrence of documented disease progression or death from any cause in the absence of progressive disease. Data was not collected due to early termination of the trial.
Time Frame: Up to 1 year
Population: Safety population. Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Part 1 and 2: Overall Survival (OS)
Description: OS is defined as the time from date of start of treatment to date of death due to any cause. Data was not collected due to early termination of the trial.
Time Frame: Up to 1 year
Population: Safety population. Part 2 was not initiated due to Sponsor's decision to terminate the trial.
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious TEAEs and SAEs were collected up to 1 year
Description: Safety Population. Only data for Part 1 has been presented as study was terminated per the sponser's decision and Part 2 was not initiated.
Arm/Group | Part 1: MT-3724 10 mcg/Kg-LEN | Part 1: MT-3724 25 mcg/Kg-LEN | Part 1: MT-3724 20 mcg/Kg-LEN | Part 2: MT-3724 50mcg/Kg-LEN
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 1/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MT-3724 10 mcg/Kg-LEN (N=3) | Part 1: MT-3724 25 mcg/Kg-LEN (N=3) | Part 1: MT-3724 20 mcg/Kg-LEN (N=3) | Part 2: MT-3724 50mcg/Kg-LEN (N=0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: MT-3724 10 mcg/Kg-LEN (N=3) | Part 1: MT-3724 25 mcg/Kg-LEN (N=3) | Part 1: MT-3724 20 mcg/Kg-LEN (N=3) | Part 2: MT-3724 50mcg/Kg-LEN (N=0)
Fatigue (General disorders) | 1 | 2 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0
Oedema peripheral (General disorders) | 0 | 3 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Left atrial enlargement (Cardiac disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Transaminase increased (Investigations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03645395/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT03645395/SAP_001.pdf